CLINICAL TRIAL: NCT02128724
Title: A CR-UK Phase I Study of BKM120 in Patients With Non-small Cell Lung Cancer (NSCLC) Receiving Thoracic Radiotherapy
Brief Title: Palliative Thoracic Radiotherapy Plus BKM120
Acronym: BKM120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Cancer Research UK (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_031; 2012-003762-40 (EudraCT Number)
Record Dates: First submitted 2014-04-16; First posted 2014-05-01 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung cancer; BKM120; Hypoxia; Misonidazole; Radiotherapy; Buparlisib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Hypoxia | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 plus radiotherapy (Experimental): Three cohorts of patients will be treated with escalating doses of oral buparlisib. The doses will be 50mg, 80mg and 100mg, once daily. Patients will be treated with buparlisib for a total of fourteen days. One week after commencing buparlisib, patients will start palliative radiotherapy treatment. Radiotherapy treatment will be delivered as 20Gy in 5 fractions over a one week period. There will be an expansion cohort at the MTD. Patients in an optional fourth cohort will take buparlisib for 4 weeks at the MTD.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — Buparlisib is a highly specific inhibitor of phosphatidylinositol 3-kinase (PI3K). Buparlisib is supplied as 10mg and 50mg hard gelatin capsules.
  Other Names: buparlisib

SUMMARY:
This study will test whether a drug called BKM120/buparlisib is a safe and effective treatment when given to lung cancer patients having radiotherapy treatment. The trial will identify which of three possible doses of buparlisib is best to give with lung radiotherapy.

DETAILED DESCRIPTION:
This study will be a single-centre, open-label, 3+3 cohort, dose escalation phase I study of the use of buparlisib in combination with thoracic radiotherapy. Patients with incurable NSCLC requiring palliative thoracic radiotherapy will be eligible for entry.

The first three cohorts of patients will be treated with escalating doses of BKM120. These patients will be treated with buparlisib for a total of fourteen days. One week after commencing buparlisib, patients will start palliative radiotherapy treatment. Radiotherapy treatment will be delivered as 20Gy in 5 fractions over a one week period. Maximum tolerated dose (MTD) will be determined and a further 6 patients will be treated at this dose. Response to buparlisib treatment will be based upon changes in tumour hypoxia and perfusion as detected by 18F-Miso PET-CT scans and perfusion CT scans respectively.

In the event that no changes are detected in tumour hypoxia or perfusion in cohorts 1-3, an optional group of patients (cohort 4) will be recruited. These patients will receive buparlisib treatment for a total of 28 days. Three weeks after commencing buparlisib, this cohort will receive palliative radiotherapy with 20Gy in 5 fractions over a one week period.

Samples from the patients will also be analysed:

Phosphorylation Status of Akt in Peripheral Blood Mononuclear Cells (PBMCs) Tumour Phosphatase and tensin homolog (PTEN) gene levels Tumour PRAS40 Levels

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histologically confirmed NSCLC of any stage
* Thoracic lesion requiring palliative radiotherapy and which has been identified on a scan within eight weeks of starting the trial.
* Male or female, age ≥ 18 years at the day of consenting to the study.
* Life expectancy of at least 16 weeks.
* ECOG performance score of 0-2.
* Patient is able to swallow and retain oral medication.
* The patient is willing to provide written informed consent and is likely to comply with the protocol for the duration of the study, and scheduled follow-up visits and examinations.
* Haematological and biochemical indices within the ranges shown below:

  * Haemoglobin (Hb) ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelet count ≥100 x 109/L
  * International Normalised Ratio (INR) ≤ 1.5
  * Potassium, calcium and Magnesium within normal range
  * ALT and AST not above normal range or ≤3.0 times ULN if liver metastases are present
  * Total serum bilirubin not above normal range, or ≤1.5 times ULN if liver metastases are present or total bilirubin ≤3.0 times ULN if the patient has well documented Gilbert's disease and absence of other contributing disease process at the time of diagnosis
  * Creatinine ≤ 1.5 x ULN
  * Fasting plasma glucose (FPG) ≤ 120mg/dL [6.7 mmol/L]

Exclusion Criteria:

* Previous chemotherapy or biological therapy within four weeks of starting study treatment.
* Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment.
* Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy.
* Treatment at the start of study treatment with any drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A4, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Presence of active uncontrolled or symptomatic CNS metastases. Patients with asymptomatic CNS metastases may participate in this trial. Any prior local treatment for CNS metastases must have been completed treatment ≥ 28 days prior to enrolment in the trial (including surgery and radiotherapy).
* Patient has poorly controlled diabetes mellitus (HbA1c > 8 %)
* Previous exposure to PI3K, mTOR, or AKT inhibitor
* Patient has a known hypersensitivity to any of the excipients of BKM120
* Previous thoracic radiotherapy treatment
* Any previous extra-thoracic radiotherapy within 28 days prior to enrolment
* Medically documented history of or active major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or risk of doing harm to others
* Patient meets the cut-off score of ≥ 12 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)
* Patient has ≥CTCAE grade 3 anxiety
* Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
* Patient has a concurrent malignancy or has had any malignancy (other than NSCLC) in the last 3 years prior to start of study treatment (with the exception of adequately treated basal or squamous cell carcinoma or cervical carcinoma in situ)
* Patient has had major surgery within 14 days of starting the study drug.
* Patient has any other concurrent severe, and/or uncontrolled medical condition that would, in the investigator's judgement contraindicate patient participation in the clinical study (e.g. chronic pancreatitis, chronic active hepatitis).
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120.
* Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.
* Patient has active cardiac disease or a history of myocardial infarction within 6 months of entering the trial, congestive heart failure ( New York Heart Association functional classification III-IV) or documented cardiomyopathy
* Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used. Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives. Women of child-bearing potential must have a negative serum pregnancy test less than 72 hours prior to initiating treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Higgins, MRCP, FRCR, D.Phil, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford, OXON, United Kingdom

REFERENCES:
- [Background] Fokas E, Im JH, Hill S, Yameen S, Stratford M, Beech J, Hackl W, Maira SM, Bernhard EJ, McKenna WG, Muschel RJ. Dual inhibition of the PI3K/mTOR pathway increases tumor radiosensitivity by normalizing tumor vasculature. Cancer Res. 2012 Jan 1;72(1):239-48. doi: 10.1158/0008-5472.CAN-11-2263. Epub 2011 Nov 22. PMID 22108822

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 50mg Buparlisib: These patients were treated with 50mg buparlisib OD for a total of fourteen days. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  BKM120: BKM120/buparlisib is a highly specific inhibitor of phosphatidylinositol 3-kinase (PI3K). BKM120 is supplied as 10mg and 50mg hard gelatin capsules.
- Cohort 2: 80mg Buparlisib: These patients were treated with 80mg buparlisib OD for a total of fourteen days. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  BKM120: BKM120/buparlisib is a highly specific inhibitor of phosphatidylinositol 3-kinase (PI3K). BKM120 is supplied as 10mg and 50mg hard gelatin capsules.
- Cohort 3: 100mg Buparlisib: These patients were treated with 100mg buparlisib OD for a total of fourteen days. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  BKM120: BKM120/buparlisib is a highly specific inhibitor of phosphatidylinositol 3-kinase (PI3K). BKM120 is supplied as 10mg and 50mg hard gelatin capsules.
- 100mg Buparlisib Expansion Cohort: These patients were treated with 100mg buparlisib OD for a total of fourteen days, after 100mg buparlisib OD was determined to be the MTD. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  BKM120: BKM120/buparlisib is a highly specific inhibitor of phosphatidylinositol 3-kinase (PI3K). BKM120 is supplied as 10mg and 50mg hard gelatin capsules.
Period: Overall Study
Arm/Group | Cohort 1: 50mg Buparlisib | Cohort 2: 80mg Buparlisib | Cohort 3: 100mg Buparlisib | 100mg Buparlisib Expansion Cohort
Started | 4 | 4 | 3 | 10
Completed | 3 | 3 | 3 | 7
Not Completed | 1 | 1 | 0 | 3
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Phase: Cohort 1: Patients treated at 50mg buparlisib once daily for a total of fourteen days for the dose escalation phase. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
- Dose Escalation Phase: Cohort 2: Patients treated at 80mg buparlisib once daily for a total of fourteen days for the dose escalation phase. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
- Dose Escalation Phase: Cohort 3: Patients treated at 100mg buparlisib once daily for a total of fourteen days for the dose escalation phase. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
- Dose Expansion Phase: Patients treated at 100mg buparlisib once daily for a total of fourteen days after the MTD had been established at 100mg buparlisib. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 | Dose Expansion Phase | Total
Number analyzed (Participants) | 4 | 4 | 3 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 64 [58 to 77] | 72 [63 to 75] | 68 [68 to 72] | 68 [52 to 78] | 69 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 8 | 14
  Male | 2 | 2 | 1 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 3 | 10 | 21
Stage of Disease IV [Count of Participants; unit: Participants] | 4 | 4 | 3 | 10 | 21
Gross tumour volume [Median (Full Range); unit: mL] | 111 [13 to 510] | 135 [29 to 204] | 54 [40 to 219] | 99 [8 to 250] | 101 [8 to 510]
Histology: Adenocarcinoma [Count of Participants; unit: Participants] | 3 | 1 | 1 | 6 | 11
Histology: Squamous cell [Count of Participants; unit: Participants] | 1 | 3 | 2 | 4 | 10
Prior Chemotherapy Treatment [Count of Participants; unit: Participants] | 2 | 2 | 1 | 7 | 12
Prior surgical treatment [Count of Participants; unit: Participants] | 0 | 0 | 0 | 6 | 6
Prior Extra Thoracic Radiotherapy Treatment [Count of Participants; unit: Participants] | 0 | 1 | 0 | 3 | 4
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Patients were clinically graded according to the ECOG performance scale based on their activity performance description (with 0 corresponding to the best outcome and 4 the worst).
  Participants
    ECOG PS Score 0 | 0 | 0 | 1 | 5 | 6
    ECOG PS Score 1 | 4 | 4 | 2 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Analysis: Number of DLTs Observed in Evaluable Patients
Description: The maximum tolerated dose (MTD) was defined as the highest dose at which no more than 1 of 6 evaluable patients or 0 of 3 evaluable patients experience a dose limiting toxicity (DLT). The study was carried out using a 3+3 dose escalation design.
  DLTs were defined per NCI CTCAE v 4.0. The following were considered DLT if they occur at any point whilst the patient is on study: 1) Any ≥ grade 3 non-haematological toxicity (excluding nausea, vomiting or diarrhoea) that requires hospital admission or which does not resolve to ≤ grade 2 within 7 consecutive days of optimal treatment. 2) Any ≥ grade 3 nausea, vomiting or diarrhoea will be considered DLT only if any of them persist for >48 hours despite maximum supportive care. 3) ≥ Grade 3 pneumonitis 4) Any ≥ Grade 4 haematological toxicity. 5) Mood deterioration from baseline. DLT will be any grade ≥3 mood change if BL score of 2. DLT will be any grade ≥2 mood change if baseline score of ≤ 1.
Time Frame: 8 weeks (10 weeks cohort 4 - this cohort was not opened)
Population: The Primary Dose Escalation analysis (the declaration of MTD) included all patients completing 14 days of buparlisib treatment and 56 days of evaluation or patients who withdrew early after experiencing DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Safety and Tolerability Analysis: Patients With Buparlisib Related Adverse Events
Description: Adverse events (AEs) and Serious Adverse Events (SAEs) were also analysed for frequency. For further details, please consult the AEs/SAEs section.
Time Frame: 8 weeks (10 weeks cohort 4 - this cohort was not opened)
Population: The safety and tolerability post-treatment analysis was based on all patients who received at least one MTD dose of buparlisib (n = 21).
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Phase: Cohort 3 and Dose Expansion Phase: Dose Escalation Phase: Cohort 3 represents patients treated at 100mg buparlisib once daily for a total of fourteen days for the dose escalation phase. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  The Dose Expansion Phase represents patients treated at 100mg buparlisib once daily for a total of fourteen days after the MTD had been established at 100mg buparlisib. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 4 | 4 | 13
Participants
  Patients with Serious Adverse Events (SAEs) | 1 | 2 | 1
  Patients with Grade >=3 Adverse Events | 1 | 2 | 5
  Patients discontinued because of AEs | 0 | 1 | 0
  Patients discontinued because of SAEs | 0 | 1 | 1

3. Secondary Outcome: Changes in 18F-Misonidazole Uptake as Detected by PET-CT Scans: Response
Description: 18F-Miso is a radiotracer that selectively accumulates in hypoxic tissues. 18F-Miso PET-CT scans are able to non-invasively image tumour hypoxia. A 18F-Miso PET-CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour hypoxia due to buparlisib treatment. For tumour hypoxia, a patient is classified as a 'responder' if there is evidence of a 10% or greater reduction in retained F-Misonidazole. Hypoxia was measured using TBRmean or TBRvolume (tumour-to-blood ratio).
Time Frame: Days -1 and 8
Population: The tumour hypoxia analysis involved all patients who had a pair of interpretable 18F-Miso PET scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 9
Participants
  Responder | 0 | 3 | 7
  Non-Responder | 3 | 0 | 2

4. Secondary Outcome: Blood Flow at Days -1 and 8 as Detected by Perfusion CT
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology due to buparlisib treatment.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: mL/100g/min
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
mL/100g/min
  pCT blood flow 1st scan | 64.2 [42 to 88.4] | 102.2 [55.8 to 106.2] | 63.9 [51.4 to 92.9]
  pCT blood flow 2nd scan | 60.2 [42.6 to 118.5] | 63.9 [51.4 to 92.9] | 64.5 [41.6 to 86.9]

5. Secondary Outcome: Tumour-to-blood Volume Ratio in 18F-Misonidazole Uptake as Detected by Day -1 and Day 8 PET-CT Scans, to Investigate if Buparlisib Alters Hypoxia
Description: 18F-Miso is a radiotracer that selectively accumulates in hypoxic tissues. 18F-Miso PET-CT scans are able to non-invasively image tumour hypoxia. A 18F-Miso PET-CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment.
  Tumour to blood volume ratio ("TBR volume") is measured by summing the number of tumour/node/metastases voxels with a value greater than or equal to 1.4.
Time Frame: Days -1 and 8
Population: The tumour hypoxia analysis involved all patients who had a pair of interpretable PET scans.
Measure: Median (Inter-Quartile Range); unit: Tumour to blood volume ratio
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 9
Tumour to blood volume ratio
  First scan | 44.4 [0.4 to 239] | 51.3 [1.3 to 99.5] | 33.1 [6.9 to 43.7]
  Second scan | 47.6 [0.4 to 233] | 42.2 [1.1 to 75.6] | 25.4 [4.9 to 42.0]

6. Secondary Outcome: Changes in Blood Flow as Detected by Perfusion CT: Response
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology due to buparlisib treatment. For tumour perfusion, a patient is classified as 'responder' if blood flow (BF) and/or blood volume (BV) is increased and/or mean transit time (MTT) is reduced from baseline measurements by more than 25%.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
Participants
  Responder | 2 | 0 | 3
  Non-Responder | 1 | 3 | 5

7. Secondary Outcome: Percentage Change in Blood Flow as Detected by Perfusion CT at Days -1 and 8
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology (blood flow) due to buparlisib treatment, and the percentage change between both scans calculated.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: % change in mL/100g/min
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
% change in mL/100g/min | 1.4 [-6.2 to 34.0] | -17.5 [-35.1 to 11.0] | -15.0 [-33.7 to 16.7]

8. Secondary Outcome: Tumour-to-blood Mean Ratio in 18F-Misonidazole Uptake as Detected by PET-CT Scans, to Investigate if Buparlisib Alters Hypoxia
Description: 18F-Miso is a radiotracer that selectively accumulates in hypoxic tissues. 18F-Miso PET-CT scans are able to non-invasively image tumour hypoxia. A 18F-Miso PET-CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour hypoxia due to buparlisib treatment.
  Hypoxia was measured using TBRmean and TBRvolume (tumour-to-blood ratio mean, tumour-to-blood ratio volume).
  TBR mean is measured by dividing all tumour/node/metastases voxels by the mean value of the descending aorta activity concentration.
Time Frame: Days -1 and 8
Population: The tumour hypoxia analysis involved all patients who had a pair of interpretable PET scans.
Measure: Median (Inter-Quartile Range); unit: Tumour to blood mean ratio
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 9
Tumour to blood mean ratio
  First scan | 1.34 [0.89 to 1.39] | 1.2 [0.94 to 1.42] | 1.23 [1.11 to 1.25]
  Second scan | 1.41 [1.03 to 1.47] | 1.07 [0.91 to 1.37] | 1.17 [1.11 to 1.25]

9. Secondary Outcome: Tumour-to-blood Volume Ratio Percentage Changes Between Day -1 and Day 8 in 18F-Misonidazole Uptake as Detected by PET-CT Scans, to Investigate if Buparlisib Alters Hypoxia
Description: 18F-Miso is a radiotracer that selectively accumulates in hypoxic tissues. 18F-Miso PET-CT scans are able to non-invasively image tumour hypoxia. A 18F-Miso PET-CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour hypoxia due to buparlisib treatment. The percentage change between the TBR volume for the 1st and 2nd scans was calculated.
  TBR volume is measured by summing the number of tumour/node/metastases voxels with a value greater than or equal to 1.4.
  Hypoxia was measured using TBRmean and TBRvolume (tumour-to-blood ratio mean, tumour-to-blood ratio volume).
Time Frame: Days -1 and 8
Population: The tumour hypoxia analysis involved all patients who had a pair of interpretable PET scans.
Measure: Median (Inter-Quartile Range); unit: % change in tumour to blood volume ratio
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 9
% change in tumour to blood volume ratio | 7.1 [-2.5 to 14.3] | -17.6 [-24.1 to 16.7] | -19.9 [-41.9 to 14.6]

10. Secondary Outcome: Percentage Changes in Blood Volume Between Day -1 and Day 8 as Detected by Perfusion CT
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology due to buparlisib treatment, and the % change between the 2 scans calculated.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: % change in mL/100g
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
% change in mL/100g | -11.1 [-27.8 to 5.0] | -25.0 [-34.7 to 4.6] | -21.2 [-46.3 to 6.2]

11. Secondary Outcome: Blood Volume at Day -1 and Day 8 as Detected by Perfusion CT
Description: as for outcome 4
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: mL/100g
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
mL/100g
  pCT first scan | 4.0 [3.6 to 9.0] | 6.5 [4.0 to 7.2] | 5.8 [4.3 to 7.5]
  pCT second scan | 3.8 [2.6 to 8.0] | 4.7 [3.0 to 6.2] | 5.6 [3.2 to 5.9]

12. Secondary Outcome: Mean Transit Time as Detected by Perfusion CT at Days -1 and 8
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology (blood flow) due to buparlisib treatment.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
seconds
  pCT first scan | 8.6 [6.3 to 11.2] | 7.8 [6.4 to 8.1] | 7.4 [6.6 to 8.0]
  pCT second scan | 6.2 [5.8 to 8.3] | 6.2 [6.1 to 10.1] | 6.7 [5.7 to 7.5]

13. Secondary Outcome: Percentage Change in Mean Transit Time as Detected by Perfusion CT at Days -1 and 8
Description: Perfusion CT is a technique used to study the vasculature within tumours and other tissues. It is non-invasive and readily incorporated into existing CT protocols using conventional contrast agents. A perfusion CT scan was conducted prior to commencing buparlisib and repeated prior to commencing radiotherapy treatment to identify changes in tumour physiology (blood flow) due to buparlisib treatment, and the % change between the 2 scans was calculated.
Time Frame: Days -1 and 8
Population: The tumour perfusion analysis involved all patients who had a pair of interpretable pCT scans.
Measure: Median (Inter-Quartile Range); unit: % change in seconds
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 8
% change in seconds | -25.9 [-27.9 to 7.9] | -3.1 [-21.89 to 24.7] | -12.6 [-17.8 to 2.0]

14. Other Pre Specified Outcome: Determine Phosphorylation Status of Akt in Peripheral Blood Mononuclear Cells (PBMCs)
Description: The levels of phospho-Akt expression in normal tissues may reflect the efficacy of BKM120. Changes in phospho-Akt expression will be monitored during the trial using PBMCs taken during the trial.
  Reductions in phospho-Akt expression of PBMC's following BKM120 treatment were to be correlated with changes observed with the functional imaging investigations; however it was not possible to draw any meaningful conclusions due to huge inter- and intra- participant variability seen on staining (no scoring was performed).
Time Frame: Baseline, days 8, 14, 28 and 56
Population: No scoring was performed, as on staining it was determined that the inter- and intra- participant variability seen would prevent any meaningful conclusions from being drawn.
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 0 | 0 | 0

15. Other Pre Specified Outcome: Measure Tumour PTEN (Phosphatase and Tensin Homolog Gene) Levels
Description: Exploratory studies aimed to correlate response to buparlisib with activation of specific molecular pathways present in the archived, diagnostic, tumour biopsy sample.
Time Frame: Archival sample taken before trial entry
Population: Where possible, tissue was obtained from trial participants' diagnostic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 2 | 3 | 4
Participants
  Positive | 1 | 3 | 3
  Negative | 1 | 0 | 1

16. Other Pre Specified Outcome: Measure Tumour PRAS40 Levels
Description: Exploratory studies will aim to correlate response to BKM120 with activation of specific molecular pathways present in the archived, diagnostic, tumour biopsy sample.
Time Frame: Archival sample taken before trial entry
Population: Where possible, tissue was obtained from the trial participants' clinical diagnostic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
Number analyzed (Participants) | 3 | 3 | 9
Participants
  Positive | 2 | 3 | 4
  Negative | 0 | 0 | 0
  Insufficient tissue | 1 | 0 | 5

ADVERSE EVENTS:
Time Frame: The Investigator monitored each patient for clinical and laboratory evidence of adverse events on a routine basis throughout the study from the point of receiving any research procedures through study completion.
Description: Participants were assessed for adverse events by site staff during their participation in the trial.
Groups:
- Dose Escalation Phase: Cohort 3 and Dose Expansion Phase: Dose Escalation Phase: Cohort 3 consisted of patients treated at 100mg buparlisib once daily for a total of fourteen days for the dose escalation phase. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
  The Dose Expansion Phase consisted of patients treated at 100mg buparlisib once daily for a total of fourteen days after the MTD had been established at 100mg buparlisib. One week after commencing buparlisib, patients started palliative radiotherapy treatment. Radiotherapy treatment was delivered as 20Gy in 5 fractions over a one week period.
Arm/Group | Dose Escalation Phase: Cohort 1 | Dose Escalation Phase: Cohort 2 | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 2/13
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase: Cohort 1 (N=4) | Dose Escalation Phase: Cohort 2 (N=4) | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase (N=13)
Lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase: Cohort 1 (N=4) | Dose Escalation Phase: Cohort 2 (N=4) | Dose Escalation Phase: Cohort 3 and Dose Expansion Phase (N=13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2)
Chest Pain (General disorders) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (5) | 10 (13)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Radiotherapy Dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Peripheral ischaemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Heterophoria (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fungating wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT02128724/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02128724/SAP_001.pdf